CLINICAL TRIAL: NCT00107484
Title: Phase II Study of Combidex in Axillary Node Staging in Breast Cancer
Brief Title: Magnetic Resonance Imaging Using Ferumoxtran-10 in Finding Metastases to the Axillary Lymph Nodes in Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Martha Wellons, Massey Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000420833; P30CA016059 (NIH); MCV-4141; NCI-7029
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2010-05-03 (Estimated); Status verified 2010-04

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — ferumoxtran-10; Magnetic Resonance Spectroscopy; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ferumoxtran-10
Procedure: magnetic resonance imaging
Procedure: sentinel lymph node biopsy

SUMMARY:
RATIONALE: Diagnostic procedures, such as magnetic resonance imaging (MRI) using ferumoxtran-10, may help find and diagnose breast cancer that may have spread to the axillary lymph nodes and may help in planning breast cancer treatment.

PURPOSE: This phase II trial is studying how well MRI using ferumoxtran-10 works in finding metastases to the axillary lymph nodes in patients with invasive breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the utility of magnetic resonance (MR) imaging using ferumoxtran-10 in identifying metastases to the axillary lymph nodes in patients with invasive breast cancer.

Secondary

* Determine the changes in MR T1 and T2 signal intensity in primary breast tumors after administration of this drug to these patients.
* Determine the potential of delayed imaging, in terms of defining tumor boundaries, in these patients.

OUTLINE: Patients receive ferumoxtran-10 IV over 25-30 minutes on day 0 in the absence of unacceptable toxicity. Patients undergo MRI of the involved breast and ipsilateral axilla on day 0 (once before and once after ferumoxtran-10 administration) and then once on day 1.

Within 3 weeks after the completion of imaging studies, patients undergo sentinel lymph node biopsy. If the sentinel node is positive for malignancy on touch prep, an axillary lymph node dissection is performed if clinically indicated.

Patients are followed at approximately 1 month after surgery.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study within 8.3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed invasive breast cancer
* Candidate for sentinel lymph node biopsy and/or axillary lymph node dissection
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count > 100,000/mm^3
* Ferritin ≤ 350 ng/mL*
* Transferrin saturation level ≤ 40%* NOTE: *Patients with lab values above these limits may be eligible provided there is no hemochromatosis by hematology consultation

Hepatic

* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Alkaline phosphatase normal
* PT normal
* Albumin normal
* No history of cirrhosis

Renal

* Creatinine normal OR
* Creatinine clearance > 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Medically stable
* No ongoing or active infection
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to ferumoxtran-10 (e.g., iron preparations, parenteral iron, parenteral dextran, parenteral iron-dextran, or parenteral iron-polysaccharide preparations)
* No history of allergic reaction to any contrast media
* No immunodeficiency that would predispose patient to a specific or non-specific mediator release
* No contraindication to MRI, including any of the following:

  * Severe claustrophobia
  * Pacemaker
  * Aneurysm clips
  * Defibrillators
  * Certain types of replacement joints
  * Other institutional contraindication to MRI
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 30 days since prior investigational agents
* More than 3 months since prior ferumoxides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2005-09; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Utility of magnetic resonance imaging using ferumoxtran-10 in identifying metastases to axillary lymph nodes | 2 years

SECONDARY OUTCOMES:
Changes in MR T1 and T2 signal intensity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Karen A. Kurdziel, MD, Study Chair — Massey Cancer Center
Locations (1):
- Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia, United States